CLINICAL TRIAL: NCT06257732
Title: Investigation of Effectiveness of Different Exercise Types, and Their Therapeutic Effect Mechanisms and the Roles of Motivational Interview in the Treatment of Non-Alcoholic Fatty Liver Disease
Brief Title: Different Exercise Modalities in the Treatment of NAFLD and Their Impact on Myokines
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeditepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBTK-MK-2022
Record Dates: First submitted 2024-01-05; First posted 2024-02-14 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-01

CONDITIONS: NAFLD; Nonalcoholic Fatty Liver Disease; Fatty Liver, Nonalcoholic; Fatty Liver
Keywords: Exercise; Myokine; HIIT; Fatmax Intensity; Resistance Exercise; Motivational Interviewing; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Motor Activity | interventions — Exercise; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control Group (No Intervention): This group will consist of individuals with liver fat accumulation under standard care and no exercise intervention will be implemented.
- Fatmax Exercise Group (Experimental): Individuals with liver fat accumulation under standard care will have their Fatmax values calculated and an exercise prescription will be designed accordingly.
  Interventions: Other: Exercise
- Fatmax Exercise and Motivational Interviewing Group (Experimental): In addition to the prescription of Fatmax exercise for individuals with liver fat accumulation under standard care, motivational interviewing principles will be applied.
  Interventions: Other: Exercise; Behavioral: Motivational Interviewing
- HIIT Group (Experimental): Individuals with liver fat accumulation under standard care will be provided with a High-Intensity Interval Training (HIIT) exercise prescription.
  Interventions: Other: Exercise
- HIIT and Motivational Interviewing Group (Experimental): In addition to formulating a High-Intensity Interval Training (HIIT) exercise prescription for individuals with liver fat accumulation under standard care, motivational interviewing principles will be applied.
  Interventions: Other: Exercise; Behavioral: Motivational Interviewing
- Resistance Exercise Group (Experimental): Individuals with liver fat accumulation under standard care will be provided with a resistance exercise prescription.
  Interventions: Other: Exercise
- Resistance Exercise and Motivational Interviewing Group (Experimental): In addition to formulating a resistance exercise prescription for individuals under standard care with liver fat accumulation, motivational interviewing principles will be applied.
  Interventions: Other: Exercise; Behavioral: Motivational Interviewing

INTERVENTIONS:
Other: Exercise — The exercise interventions in this study include High-Intensity Interval Training (HIIT), involving brief bursts of intense exercise; Resistance Exercise, focusing on strength and muscle endurance; and Fatmax Exercise, tailored to optimize fat oxidation during aerobic activity.
  Arms: Fatmax Exercise Group; Fatmax Exercise and Motivational Interviewing Group; HIIT Group; HIIT and Motivational Interviewing Group; Resistance Exercise Group; Resistance Exercise and Motivational Interviewing Group
Behavioral: Motivational Interviewing — Motivational Interviewing will be employed as a counseling technique to elicit behavior change by fostering collaborative and empathetic conversations, enhancing motivation for positive lifestyle modifications in individuals with liver fat accumulation.
  Arms: Fatmax Exercise and Motivational Interviewing Group; HIIT and Motivational Interviewing Group; Resistance Exercise and Motivational Interviewing Group

SUMMARY:
The goal of this 12-week clinical trial is to investigate the effectiveness of different exercise types in treating Non-Alcoholic Fatty Liver Disease (NAFLD) and to explore their impact on myokine levels associated with lipid metabolism. The main questions it aims to answer are:

1. How does the type and dose of exercise affect the treatment of NAFLD?
2. What is the influence of exercise interventions in NAFLD treatment on myokine levels related to lipid metabolism?
3. How does motivational interviewing contribute to lifestyle modification in the treatment of NAFLD?

Participants in this study will engage in assigned exercise routines randomly, including HIIT, resistance training, or FATmax exercises. Additionally, motivational interviewing techniques will be employed to assess their impact on lifestyle changes. Researchers will compare the outcomes among the different exercise groups, along with a control group receiving only standard care for NAFLD. This comparison aims to determine the respective effects of these interventions on both NAFLD and associated myokine levels.

ELIGIBILITY:
Inclusion Criteria:

* Have received a diagnosis of Non-Alcoholic Fatty Liver Disease (NAFLD)
* Age between 25 and 50 years old
* Use of smartphone
* Fall into category A or B according to the American Heart Association Risk Assessment Criteria

Exclusion Criteria:

* Viral hepatitis
* Excessive alcohol consumption (more than 30 grams per day for men and more than 20 grams per day for women)
* Use of specific medications: amiodarone, corticosteroids, methotrexate, tamoxifen, synthetic estrogen, valproic acid, intravenous tetracycline, and highly active antiretroviral drugs
* Presence of accompanying chronic diseases such as Wilson's disease, hemochromatosis, and celiac disease
* Liver storage diseases
* Cancer
* Cirrhosis
* Advanced changes in liver ultrasonography evaluations, such as fibrosis
* Presence of other chronic diseases (kidney failure, heart failure, atherosclerotic heart disease, hypertension, arrhythmia disorders)
* BMI greater than 40 kg/m²
* History of surgery or trauma in the last 6 months
* Orthopedic and/or neurological impairment
* Health problems that may hinder participation in the exercise program
* Regular and continuous participation in sports or exercise at least 3 times a week for the past 3 years
* Family history of coronary artery disease (coronary artery disease before the age of 45 in male first-degree relatives and other male relatives, or before the age of 65 in female first-degree relatives and other female relatives)
* Presence of specific symptoms during medical history or physical examination: chest pain radiating to the neck, jaw, or arm, shortness of breath during rest or physical activity, dizziness, fainting, orthopnea or paroxysmal nocturnal dyspnea, ankle edema, palpitations or tachycardia, intermittent claudication, heart murmur, unexplained excessive fatigue
* Fall into category C or D according to the American Heart Association Risk Assessment Criteria

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in the liver steatosis grade | 12-week
  Changes in the level of liver fat accumulation in radiological abdominal ultrasonography (USG) will be observed. The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.

SECONDARY OUTCOMES:
ALT | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
AST | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
GGT | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
Free fatty acids | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
Triglycerides | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
HDL | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
LDL | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
Total cholesterol | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
CRP | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
ESR | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
Changes in body weight | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
Changes in lean body mass | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
Changes in body fat percentage | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
Changes in body mass index | 12-week
  The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
Changes in waist-to-hip ratio | 12-week
  The waist and hip measurements will be taken twice with a tape measure. The results will be aggregated to arrive at one reported value as a waist-to-hip ratio. This is calculated as waist measurement divided by hip measurement (W⁄H). The difference between the values obtained at the beginning of the study and those measured after completing the program will be evaluated. Data collected at the beginning and end of the study will be compared.
Changes in peak oxygen consumption | 12-week
  At the beginning, every 4 weeks, and at the end of the study, peak oxygen consumption measurement will be conducted through the cardiopulmonary exercise test. Data collected at the beginning and end of the study will be compared.
Changes in peak heart rate | 12-week
  At the beginning, every 4 weeks, and at the end of the study, peak heart rate measurement will be conducted through the cardiopulmonary exercise test. Data collected at the beginning and end of the study will be compared.
Changes in anaerobic threshold | 12-week
  At the beginning, every 4 weeks, and at the end of the study, anaerobic threshold measurements will be conducted through the cardiopulmonary exercise test. Data collected at the beginning and end of the study will be compared.
Changes in basal metabolic rate | 12-week
  Basal metabolic rate measurements will be conducted twice using an indirect calorimeter, once at the beginning and once at the end of the study. Data collected at the beginning and end of the study will be compared.
Changes in muscle strength analysis results | 12-week
  At the beginning and end of the study, the maximum isometric contraction strength of the hand and forearm muscles will be measured using a hand dynamometer. Data collected at the beginning and end of the study will be compared.
Changes in The 5 Times Sit-to-Stand Test results | 12-week
  The 5 Times Sit-to-Stand Test will be administered as a balance test. Data collected at the beginning and end of the study will be compared.
Changes in Single Leg Standing Test results | 12-week
  The Single Leg Standing Test will be administered as a balance test. Data collected at the beginning and end of the study will be compared.
Changes in FATmax levels | 12-week
  At the beginning and end of the study, participants' FATmax levels will be determined through the FATmax test. Data collected at the beginning and end of the study will be compared.
Changes in Healthy Lifestyle Habits Scale II scores | 12-week
  At the beginning and end of the study, a total of two administrations of the questionnaires will be conducted. Data collected at the beginning and end of the study will be compared.
Changes in Short Form Survey (SF-36) scores | 12-week
  At the beginning and end of the study, a total of two administrations of the questionnaires will be conducted. Data collected at the beginning and end of the study will be compared.
Changes in Beck Depression Scale scores | 12-week
  At the beginning and end of the study, a total of two administrations of the questionnaires will be conducted. Data collected at the beginning and end of the study will be compared.
Changes in Pittsburgh Sleep Quality Index scores | 12-week
  At the beginning and end of the study, a total of two administrations of the questionnaires will be conducted. Data collected at the beginning and end of the study will be compared.
Changes in the serum levels of myokines | 12-week
  Serum samples will be obtained twice, at the beginning and end of the study. Musclin, myonectin, and myostatin levels will be measured using ELISA, while measurements of BAIBA will be conducted using Liquid Chromatography Spectrometry. Data collected at the beginning and end of the study will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No